CLINICAL TRIAL: NCT00576368
Title: An Open Therapeutic Project to Confirm the Efficacy Tolerability and Safety Profile of Lantus in Everyday Medical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_5007
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — The physician will be guided by the prescribing information outlined in the summary of product characteristics. The administration will be done by once daily subcutaneous injection.

SUMMARY:
The objective of this survey on this registered product is to confirm the efficacy, and safety profile of Lantus in every day medical practice. This program will also help to obtain information about the use of the insulin titration regimen and handling of the Lantus insulin analogue.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed diabetics and existing diabetics uncontrolled on other anti-diabetic therapy, where treatment with basal insulin is required to control hyperglycaemia, and who the treating investigator considers may benefit from the treatment with Lantus, could enter in this program.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4464 (Actual)
Dates: Start 2003-06; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Glycemic status (Fasting Blood Glucose, Fasting Plasma Glucose, and HbA1C as done in routine medical practice) | at least 3months

CONTACTS AND LOCATIONS:
Overall Officials: E Hens, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Brussels, Belgium